CLINICAL TRIAL: NCT06739213
Title: SYHA1813 vs Investigators' Choice as Treatment for Recurrent or Progressive High-Grade Meningioma: A Randomized, Controlled, Multicenter, Phase II Study
Brief Title: A Phase II Study of SYHA1813 for Recurrent or Progressive High-Grade Meningioma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYHA1814-004
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Recurrent or Progressive High Grade Meningioma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, open-label, multicenter, Phase II clinical trail, randomized 1:1 to receive either SYHA1813 (experimental group) or investigators' choice (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): SYHA1813
  Interventions: Drug: SYHA1813
- Control group (Active Comparator): Investigator's Choice Treatment
  Interventions: Drug: Investigator's Choice Treatment

INTERVENTIONS:
Drug: SYHA1813 — The starting dose of SYHA1813 is 20mg QD
  Arms: Experimental group
Drug: Investigator's Choice Treatment — Investigator's Choice Treatment
  Arms: Control group

SUMMARY:
This is a randomized, controlled, open-label, multicenter, Phase II clinical study designed to evaluate the efficacy and safety of SYHA1813 compared to investigators' choice in participants with recurrent or progressive high-grade meningioma.

DETAILED DESCRIPTION:
A total of 56 participants with recurrent or progressive high-grade meningioma who are not eligible for local therapy will be enrolled. Participants will be randomized 1:1 to receive either SYHA1813 (experimental group) or investigators' choice (control group). The primary endpoint is the 6-month progression-free survival (PFS) rate assessed by investigators using the Response Assessment in Neuro-Oncology Working Group（ RANO criteria） for meningioma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >= 18 years;
2. Histologically confirmed WHO grade II/III meningioma (WHO CNS 5th)
3. There is at least one measurable lesion in the baseline period (RANO-meningioma);
4. KPS≥60;
5. The expected survival time is >=3 months;
6. The organ function level and related laboratory indicators must meet requirements (no blood transfusion within 2 weeks):
7. Female participants of childbearing potential must have a negative the blood pregnancy test results of within 7 days prior to randomization and agree to use reliable and effective contraception during the study treatment period and for at least 3 months after the last study treatment (or as required by the drug's instructions). Male participants with partners of childbearing potential must agree to use reliable and effective contraception during the study treatment period and for at least 3 months after the last study treatment (or as required by the drug's instructions).

Exclusion Criteria:

1. Patients who are known or suspected to be allergic to the test drug or its components;
2. Meets one of the following conditions: patients with brainstem involvement; patients with severe brain herniation or at risk of brain herniation; patients with extracranial metastasis during the screening period.
3. A history of any other malignant tumors within 3 years (except for effectively controlled skin basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer or cured carcinoma in situ);
4. Use of glucocorticoids at an equivalent dose exceeding 5mg of dexamethasone within 7 days prior to randomization.
5. The toxicity of previous anti-tumor treatments has not recovered to Grade1(including brain edema after radiotherapy), with the exception of hair loss, uncomplicated laboratory abnormalities that do not require medical intervention, and other adverse reactions deemed by the investigator not to affect the safety of the study medication.;
6. Use of a strong CYP3A4 inhibitor within 14 days prior to randomization or ongoing use of such inhibitors.
7. Current use of warfarin or other oral anticoagulants (except for low-dose anticoagulants used to maintain central venous access or prevent deep vein thrombosis).
8. Inability to undergo contrast-enhanced MRI
9. Patients with evidence of bleeding tendency or medical history within 2 moths
10. Urine protein ≥ 2+, and 24-hour urine protein quantitative ≥ 1.0g/24h;
11. Human immunodeficiency virus (HIV) antibody positive; active hepatitis C (anti-HCV antibody positive and HCV RNA test positive); active hepatitis B (HBV DNA test for HBsAg is positive and HBV DNA is equal to or higher than 2×10^3 IU/ml));
12. The subject has poorly healed wounds, ulcers or fractures;
13. Presence of a severe chronic or active infection (including tuberculosis and other infections).requiring intravenous antibiotic, antifungal, or antiviral treatment within 14 days prior to randomization
14. Other severe systemic diseases, including but not limited to uncontrolled diabetes, kidney disease requiring dialysis, severe liver disease (Child-Pugh class B or C), acute pancreatitis, etc.
15. Subjects with clinically significant cardiovascular and cerebrovascular diseases.
16. Underwent major organ surgery within 28 days prior to randomization (excluding biopsy procedures).
17. Received chemotherapy (including temozolomide), targeted therapy, immunotherapy, hormone therapy, or other antitumor treatments within 28 days prior to randomization; or used any NMPA-approved traditional Chinese medicine or patent Chinese medicine with anticancer activity within 14 days prior to randomization (regardless of cancer type).
18. Subjects with dysphagia or known drug absorption disorders.
19. Pregnant or lactating women.
20. Presence of other conditions that may interfere with the participant's ability to comply with the study procedures or that may not allow the participant to derive the maximum benefit from the study, or that may affect the study outcomes, such as a history of psychiatric disorders, drug or substance abuse, or any other clinically significant disease or condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
the Progression-free survival (PFS) at 6-month（PFS-6）as evaluated by investigator (RANO-meningioma) | Up to approximately 3years

SECONDARY OUTCOMES:
Progression-free survival (PFS) as evaluated by INV (RANO-meningioma) | Up to approximately 3years
Objective response rate (ORR) as evaluated by INV (RANO-meningioma) | Up to approximately 3years
Disease control rate (DCR) as evaluated by INV (RANO-meningioma) | Up to approximately 3years
Overall survival (OS) | Up to approximately 3years
Frequency and severity of TEAE and SAE | Up to approximately 3years
Maximum Plasma Concentration of SYHA1813 (Cmax) | Up to approximately 3years
The scores of the 30-item European Organisation for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) | Up to approximately 3years
  The EOTCT QLQ-C30 is designed to measure the health-related quality of life (HRQoL) across different cancer types and stages. It has demonstrated good evidence of content validity for assessing functional health, symptom burden, and health-related quality of life in patients with localized to advanced cancer. The questionnaire comprises 30 items that are combined to form five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea/vomiting), and six single items (appetite loss, diarrhea, constipation, dyspnea, insomnia, and financial difficulties), as well as a global health status/quality of life scale. The global health status scale is scored on a 7-point scale, while the other items are scored on a 4-point scale. Higher scores indicate a higher level of response.
The scores of the 20-item EORTC QLQ for Brain Neoplasm (-BN20) | Up to approximately 3years
  The EORTC QLQ-BN20 is a 20-item questionnaire specifically designed for assessing the health-related quality of life (HRQOL) and symptoms in patients with brain cancer, including both primary brain tumors and brain metastases. Within the EORTC framework, there is a distinction between functional scales (e.g., "Emotional Functioning") and symptom scales (e.g., "Pain"). High scores on functional scales indicate better functioning, while high scores on symptom scales indicate a greater symptom burden.
The score of The Neurologic Assessment in Neuro-Oncology (NANO) scale | Up to approximately 3years
  The NANO scale evaluates 9 major domains of neurologic function that are most relevant to patients with supratentorial, infratentorial, and brainstem tumors, including gait, strength, upper extremity ataxia, sensation, visual fields, facial strength, language, level of consciousness, and behavior. As designed, the gait domain includes assessment of lower extremity ataxia. Each domain is subdivided into 3 or 4 levels of function with scores based on discrete quantifiable measures. Thus, levels of function for each domain range from 0 to 2 or 0 to 3. A score of 0 indicates normal function, while the highest score indicates the most severe level of deficit for that domain. Levels of function are distinguished by significant and measurable differences in order to avoid misinterpretation of subtle or nonspecific changes.

IPD SHARING:
Plan to Share IPD: No